CLINICAL TRIAL: NCT00201227
Title: Using Learning Teams for Reflective Adaptation
Brief Title: Trial to Enhance Adherence to Multiple Guidelines
Acronym: ULTRA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Medicine and Dentistry of New Jersey (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: Rutgers, The State University of New Jersey (Other)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: 278; R01HL070800 (NIH)
Record Dates: First submitted 2005-09-16; First posted 2005-09-20 (Estimated); Last update posted 2017-07-11 (Actual); Status verified 2015-10

CONDITIONS: Asthma; Cardiovascular Diseases; Atherosclerosis; Diabetes Mellitus; Heart Diseases; Hypertension; Lung Diseases
MeSH Terms: conditions — Asthma; Cardiovascular Diseases; Atherosclerosis; Diabetes Mellitus; Heart Diseases; Hypertension; Lung Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Practice Change (Experimental): Enhancement of primary care practice performance and practice guideline adherence
  Interventions: Other: practice guideline adherence
- Control (No Intervention): Usual care

INTERVENTIONS:
Other: practice guideline adherence — Project facilitator assist primary care practice clinicians and staff work in effective quality improvement teams through the use of facilitated collaborative meetings.
  Arms: Practice Change

SUMMARY:
To evaluate whether the innovative multimethod assessment process/participatory quality improvement (MAP/PQI) intervention increases adherence to multiple cardiorespiratory guidelines in primary care practice.

DETAILED DESCRIPTION:
BACKGROUND:

Because of its ongoing access to the majority of the U.S. population, the primary care setting has great potential for preventing and managing cardiorespiratory illness. However, due to their broad focus and competing demands, primary care practices often fail to translate evidence-based guidelines into practice. Based on more than 10 years of practice-based observational and intervention research, the investigators have developed a multimethod assessment process (MAP) for understanding the unique barriers, opportunities and complexity of diverse primary care practice settings. MAP has been used to inform a practice-individualized intervention that resulted in sustained increases of evidence-based guidelines for clinical preventive service delivery. They integrated a participatory quality improvement (PQI) process that involves patients, office staff, and physicians with MAP (MAP/PQI) to enhance and promote ongoing practice-specific quality improvement.

The study is in response to a Request for Applications on "Trials Assessing Innovative Strategies to Improve Clinical Practice Through Guidelines in Heart, Lung and Blood Diseases".

DESIGN NARRATIVE:

This study will evaluate whether the innovative MAP/PQI intervention increases adherence to multiple cardiorespiratory guidelines in primary care practice. A group randomized clinical trial of 60 primary care practices representing diverse patient populations and payment systems will be conducted. After a 2-year follow-up, the control group will cross-over to a refined delayed intervention. MAP at each practice will identify features that foster and/or impede adherence to screening and treatment guidelines for multiple cardiorespiratory diseases among the competing demands of practices. PQI will then engage clinicians, staff, and patients in implementing tailored improvements that target the whole practice and simultaneously focus on changes that affect multiple guidelines. Rates of adherence to multiple guidelines will be compared for intervention and control practices. A comparative case study process analysis will identify features associated with success. The major outcome is adherence to a select group of guidelines addressing: hypertension (chronic disease,) asthma (cyclic disease), diabetes (chronic with multiple co-morbidities), smoking (simple screening) and cholesterol (complicated). The conceptual framework is well developed by the authors with significant prior work in this area. These insights will be incorporated into a refined intervention for the control group (delayed intervention), and evaluated in a pre/post design. Tailoring MAP/PQI to unique practice characteristics is likely to result in sustained increases in adherence to cardiorespiratory guidelines. The intervention will be translatable into ongoing implementations of evidence-based guidelines in the primary care setting where the majority of Americans receive their medical care.

ELIGIBILITY:
No eligibility criteria - study subjects are medical practices, so criteria are for clinicians and staff working within these practices.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2002-09; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
practice adherence to diabetes guidelines | baseline, 1 year, 2 year, 3 year

SECONDARY OUTCOMES:
practice adherence to hypertension guideline | baseline, 1 year, 2 year, 3 year
practice adherence to asthma guidelines | baseline, 1 year, 2 year, 3 year
practice adherence to cholesterol screening guidelines | baseline, 1 year, 2 year, 3 year
practice adherence to tobacco history taking guidelines | baseline, 1 year, 2 year, 3 year

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin F Crabtree, Principal Investigator — Univ of Med/Dent/NJ-R W Johnson Medical School

REFERENCES:
- [Background] Stroebel CK, McDaniel RR Jr, Crabtree BF, Miller WL, Nutting PA, Stange KC. How complexity science can inform a reflective process for improvement in primary care practices. Jt Comm J Qual Patient Saf. 2005 Aug;31(8):438-46. doi: 10.1016/s1553-7250(05)31057-9. PMID 16156191
- [Background] Crosson JC, Stroebel C, Scott JG, Stello B, Crabtree BF. Implementing an electronic medical record in a family medicine practice: communication, decision making, and conflict. Ann Fam Med. 2005 Jul-Aug;3(4):307-11. doi: 10.1370/afm.326. PMID 16046562
- [Background] Cohen D, McDaniel RR Jr, Crabtree BF, Ruhe MC, Weyer SM, Tallia A, Miller WL, Goodwin MA, Nutting P, Solberg LI, Zyzanski SJ, Jaen CR, Gilchrist V, Stange KC. A practice change model for quality improvement in primary care practice. J Healthc Manag. 2004 May-Jun;49(3):155-68; discussion 169-70. PMID 15190858
- [Background] Ohman-Strickland PA, Orzano AJ, Hudson SV, Solberg LI, DiCiccio-Bloom B, O'Malley D, Tallia AF, Balasubramanian BA, Crabtree BF. Quality of diabetes care in family medicine practices: influence of nurse-practitioners and physician's assistants. Ann Fam Med. 2008 Jan-Feb;6(1):14-22. doi: 10.1370/afm.758. PMID 18195310
- [Background] Strickland PA, Crabtree BF. Modelling effectiveness of internally heterogeneous organizations in the presence of survey non-response: an application to the ULTRA study. Stat Med. 2007 Apr 15;26(8):1702-11. doi: 10.1002/sim.2794. PMID 17211824
- [Background] Hudson SV, Harris-Haywood S, Stange KC, Orzano AJ, Crabtree BF. Recruiting minority primary care practices into practice-based research. Med Care. 2006 Jul;44(7):696-700. doi: 10.1097/01.mlr.0000215818.38729.81. PMID 16799365
- [Background] Crosson JC, Ohman-Strickland PA, Hahn KA, DiCicco-Bloom B, Shaw E, Orzano AJ, Crabtree BF. Electronic medical records and diabetes quality of care: results from a sample of family medicine practices. Ann Fam Med. 2007 May-Jun;5(3):209-15. doi: 10.1370/afm.696. PMID 17548848
- [Background] Hudson SV, Ohman-Strickland P, Cunningham R, Ferrante JM, Hahn K, Crabtree BF. The effects of teamwork and system support on colorectal cancer screening in primary care practices. Cancer Detect Prev. 2007;31(5):417-23. doi: 10.1016/j.cdp.2007.08.004. Epub 2007 Nov 26. PMID 18031947
- [Background] Ohman-Strickland PA, John Orzano A, Nutting PA, Perry Dickinson W, Scott-Cawiezell J, Hahn K, Gibel M, Crabtree BF. Measuring organizational attributes of primary care practices: development of a new instrument. Health Serv Res. 2007 Jun;42(3 Pt 1):1257-73. doi: 10.1111/j.1475-6773.2006.00644.x. PMID 17489913
- [Background] Hahn KA, Strickland PA, Hamilton JL, Scott JG, Nazareth TA, Crabtree BF. Hyperlipidemia guideline adherence and association with patient gender. J Womens Health (Larchmt). 2006 Nov;15(9):1009-13. doi: 10.1089/jwh.2006.15.1009. PMID 17125419
- [Background] Ferrante JM, Ohman-Strickland P, Hudson SV, Hahn KA, Scott JG, Crabtree BF. Colorectal cancer screening among obese versus non-obese patients in primary care practices. Cancer Detect Prev. 2006;30(5):459-65. doi: 10.1016/j.cdp.2006.09.003. Epub 2006 Oct 25. PMID 17067753